CLINICAL TRIAL: NCT04258072
Title: Phase 1b Study of Vactosertib (TEW-7197) in Combination With Nal-IRI／FL in Patients With Metastatic Pancreatic Ductal Adenocarcinoma Who Have Failed First-Line Gemcitabine／Nab-Paclitaxel
Brief Title: Vactosertib With Nal-IRI/FL in Metastatic Pancreatic Ductal Adenocarcinoma.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, M.D., PhD,Principal Investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10-054
Record Dates: First submitted 2020-01-21; First posted 2020-02-06 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — vactosertib

STUDY DESIGN:
Intervention Model Description: * Vactosertib* 100-300 mg bid for 5 days
  * Liposomal Irinotecan (Onivyde) 70mg/m2 on D1
  * LV 200mg/m2 IV bolus on D1
  * 5-FU 2400mg/m2 CIV over 46 hours on D1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label,single arm (Experimental): Vactosertib* 100-300 mg bid for 5 days + Liposomal Irinotecan (Onivyde) 70mg/m2 + LV 200mg/m2 IV bolus + 5-FU 2400mg/m2 CIV over 46 hours
  Interventions: Drug: Vactosertib

INTERVENTIONS:
Drug: Vactosertib — Vactosertib: 50-mg white round film-coated tablets containing excipients (lactose monohydrate Fastflo 316, microcrystalline cellulose Avicel PH 102, crospovidone Kollidon CL-F, povidone Kollidon 30, magnesium stearate, opadry white) and active pharmaceutical ingredient (N-((4-([1,2,4]triazolo[1,5-a]pyridin-6-yl)-5-(6-methylpyridin-2-yl)-1H-imidazol-2-yl)methyl)-2-fluoroaniline), 10% (w/w) of total weight
  Other Names: TEW-7197

SUMMARY:
To determine recommended phase 2 dose and to evaluate the safety of vactosertib in combination with nal-IRI/FL in patients with metastatic pancreatic ductal adenocarcinoma (PDAC) who have failed first-line gemcitabine and nab-paclitaxel

DETAILED DESCRIPTION:
* Number of patients : Total 24 patients (6-12 patients in phase 1 part and 12 patients in expansion cohort )
* Treatment :

  * Vactosertib* 100-300 mg bid for 5 days
  * Liposomal Irinotecan (Onivyde) 70mg/m2 on D1
  * LV 200mg/m2 IV bolus on D1
  * 5-FU 2400mg/m2 CIV over 46 hours on D1

    * Vactosertib will be kindly provided by MedPacto.
* Disease evaluation: Tumor assessment will be conducted at screening and before Day 1 of every third cycle starting with Cycle 4
* Period : Approximately 24 months from the date of Institutional Review Board (IRB) approval
* Primary endpoint : To determine recommended phase 2 dose and to evaluate the safety of vactosertib in combination with nal-IRI/FL in patients with metastatic pancreatic ductal adenocarcinoma (PDAC) who have failed first-line gemcitabine and nab-paclitaxel
* Secondary endpoint :

  * Progression-Free Survival (PFS) (RECIST 1.1 criteria)
  * Overall Survival (OS)
  * Objective Response Rate (ORR) (RECIST 1.1 criteria)
  * Disease Control Rate (DCR) (RECIST 1.1 criteria)
* Exploratory endpoint

  * Pharmacokinetic assessment: before treatment, post treatment 1.5h, 4.5h, and 8hPharmacodynamic assessment: to evaluate changes in the amount of p-SMAD in PBMC.
  * Biomarker analysis in pre-treated and post-treated tumor samples

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are males or females ≥ 19 years of age
2. Subjects who have the following history of first-line gemcitabine-based chemotherapy among patients with cytologically or histologically proven metastatic pancreatic ductal adenocarcinoma
3. Subjects who can give written informed consent for participation in this trial after receiving explanations of this trial
4. Subjects who have the following laboratory test values:

   * bilirubin ≤ 1.5 x ULN (upper limit of normal)
   * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 x ULN
   * serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 40 mL/min (Cockcroft-Gault)
   * partial thromboplastin time (aPTT) ≤ 1.5 x ULN
   * absolute neutrophil count (ANC) ≥ 1,500 cells/µL
   * platelet count ≥ 100,000/µL
   * hemoglobin ≥ 9.0 g/dL
5. Subjects who have at least a 12-week life expectancy at the Investigator's discretion
6. Subjects who have Eastern Cooperative Oncology Group (ECOG)Performance Status 0-1

Exclusion Criteria:

1. Subjects who were treated with surgery, radiotherapy, chemotherapy or investigational therapy within 2 weeks (note: placement of biliary stent is allowed)
2. Subjects who have uncontrolled CNS metastases (patients who require steroids should be on a stable or decreasing dose for at least 2 weeks)
3. Subjects who have any contraindications for 5-FU, leucovorin, or nal-IRI
4. Subjects who have moderate or severe cardiovascular disease

   * Subjects who have myocardial infarction, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension within 6 months before screening
   * Subjects who have major abnormalities at the Investigator's discretion based on electrocardiogram (ECG)and Doppler ECHO results at screening or within 14 days before screening
   * Subjects who have increase in brain natriuretic peptide (BNP) or increase in troponin (over 99th percentile upper reference limit) at Screening (based on the normal range of relevant study center)
   * Subjects who have risk factors for ascending aortic aneurysm such as genetic disorder and trauma and risk factors for aortic stenosis
   * Subjects who have a history of heart or aorta surgery
5. Subjects who have clinically significant gastrointestinal bleeding within 4 weeks before screening
6. Subjects who have a known history or suspected hypersensitivity to any excipients of the investigational product or combination drug(s)
7. Subjects who have received prior treatment targeting the signaling pathway of TGF-β
8. Subjects who have a disease or condition that affects the mechanism of the investigational product, or are currently using or planning to use:

   * Drugs that are exclusively or primarily eliminated by cytochrome P-450 isozyme (CYP) including CYP1A2, CYP2B6, or CYP3A4
   * Drugs that are exclusively or primarily eliminated by UDP glucuronyltransferase (UGT) 1A1 (UGT1A1)
   * Drugs that are substrates for the drug transporter multidrug resistance protein 1 (MDR1) have a narrow therapeutic window or are strong inhibitors of drug transporter MDR1
   * Drugs that are strong inhibitors or inducers of CYP2D6 or CYP3A4
9. Subjects who are unable to swallow tablets
10. Subjects who have a history of or are suspected of drug abuse
11. Female subjects of child-bearing potential who have a positive result on a pregnancy test at screening or are unable to agree to use an effective barrier method of birth control to avoid pregnancy during the study period (e.g., sterilization, intrauterine contraceptive device, combination of oral contraception and barrier contraception, combination of other hormone delivery systems and barrier contraception, contraceptive cream, combination of cream, jelly, or form and diaphragm or condom)
12. Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study
13. Subjects who were treated with other investigational products within 28 days before screening or within a period shorter than 5-timesthe half-life of the investigational product

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided